CLINICAL TRIAL: NCT03497624
Title: ALCMI-006: A Prospective Biospecimen Collection Study From Patients With ROS1-Fusion Positive Tumors
Status: Completed | Type: Observational
Sponsor: Addario Lung Cancer Medical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ALCMI-006
Record Dates: First submitted 2018-03-20; First posted 2018-04-13 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: ROS1-fusion Positive Tumor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The tumor tissue will be used to develop up to 24 PDX models for ROS1-fusion driven cancers to be used for research purposes only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biospecimens collection — Collection of tumor tissue when a participant is having a clinically-indicated biopsy or surgery for their ROS1-fusion cancer.

SUMMARY:
Patient Derived Xenografts (PDXs) are models to study tumor growth, response to anti-cancer therapies, and resistance to anti-cancer therapies. The purpose of this study is to develop up to 24 PDX models for ROS1-fusion driven cancers to be used for research purposes only. That is, these patient derived PDX models will have no immediate benefit to the patient from whom the tumor specimen was obtained. Rather, these PDX models will be used to inform the study of ROS1-fusion driven cancers at large.

DETAILED DESCRIPTION:
ROS1-fusions occur in several cancer types such as non-small cell lung cancer, gastric cancer, ovarian cancer, glioblastoma, cholangiocarcinoma and melanoma. In each of these cancers, ROS1-fusions account for a small sliver of the pie, accounting for 1-2% of all diagnoses, forming a relatively rare molecular subset of cancer. The Addario Lung Cancer Medical Institute (ALCMI) would like to focus on this under-studied rare molecular subset of cancer to understand how cancer begins and spreads in these tumors, how these tumors respond to treatment and what happens when tumors stop responding to treatment. Therefore, in collaboration with cancer patients whose tumors have ROS1-fusions (known as the "ROS1ders"), we are studying ROS1-fusions across all cancer types.

Patient Derived Xenografts (PDXs) are models to study cancer. These models are developed by injecting a fresh piece of tumor specimen from a patient into a special type of mouse, which then acts as 'host' to allow the tumor to grow. Peer-reviewed and published experimental studies have shown that PDX models can maintain features similar to the original tumor from the patient. PDX models can be used to study tumor growth, response to anti-cancer therapies, and resistance to anti-cancer therapies.

The purpose of this study is to develop up to 24 PDX models for ROS1-fusion driven cancers to be used for research purposes only. That is, these patient derived PDX models will have no immediate benefit to the patient from whom the tumor specimen was obtained. Rather, these PDX models will be used to inform the study of ROS1-fusion driven cancers at large.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female greater than 18 years of age at the time of consent.
2. Confirmed diagnosis of ROS1-fusion positive tumor via IHC, FISH and/or NGS.
3. A clinically-indicated procedure (required by the patient's treating physician) scheduled no more than 30 calendar days from date of consent.
4. A minimum of 21 calendar days between the last dose of systemic therapy and the clinically-indicated procedure.
5. A minimum of 42 hours between the last dose of a tyrosine kinase inhibitor (TKI) and the time of the clinically-indicated procedure.
6. Willingness to undergo all study collection procedures and follow up.
7. Provision of written informed consent by the patient.
8. Able to communicate (read, write and speak) in English.
9. Clinically-indicated procedure to be performed within the US (including Alaska, Hawaii and Puerto Rico), Canada, England, or Israel.

Exclusion Criteria:

1. Less than 18 years of age at time of consent.
2. No confirmed diagnosis of ROS1-fusion positive tumor via IHC, FISH and/or NGS.
3. A biopsy or surgical procedure not scheduled for clinical/diagnostic purposes.
4. A clinically-indicated procedure scheduled more than 30 calendar days from the date of consent.
5. Receipt of systemic therapy less than 21 days from the time of the clinically-indicated procedure.
6. Receipt of tyrosine kinase inhibitor less than 42 hours from the time of the clinically-indicated procedure.
7. Unwilling to undergo all study collection procedures and follow up.
8. Unable or unwilling to provide consent.
9. Unable to communicate in English.
10. Clinically-indicated procedure not scheduled within the US, Canada, England, or Israel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with a ROS1-fusion positive cancer.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
The primary objective is to develop a unique cohort of PDX models for ROS1-fusion driven cancers as a resource to the research community. | 1 year
  Successful generation of at least ten (10), but no more than twenty-four (24), ROS1-fusion PDX models with full characterization including whole exome sequencing (WES) and RNA sequencing. Models can be used as a resource for clinical and translational research to understand mechanisms of resistance and develop new therapies.

SECONDARY OUTCOMES:
The secondary/exploratory objectives are to enhance scientific knowledge of how to diagnose and treat ROS1-fusion driven cancers. | 24 months
  These models will be made available to researchers to enhance scientific knowledge of how to diagnose and treat ROS1-fusion driven cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lovly, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- ALCMI, San Carlos, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined at a future date.